CLINICAL TRIAL: NCT01507662
Title: Patient Activation After DXA Result Notification
Acronym: PAADRN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fredric D Wolinsky (Other)
Collaborators: University of Alabama at Birmingham (Other); Kaiser Permanente (Other); University of Toronto (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Fredric D Wolinsky, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201107758
Record Dates: First submitted 2011-12-08; First posted 2012-01-11 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Osteoporosis; Bone Diseases, Metabolic
Keywords: Bone Density; Absorptiometry, Photon; Osteoporosis; Bone, Diseases, Metabolic; Patient Education as Topic; Fractures, Bone/Prevention and Control
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMD Result Letter and Brochure (Experimental): Patients who receive the intervention - BMD result letter with brochure.
  Interventions: Behavioral: Bone Mineral Density Result Letter and Bone Health Brochure
- Control (No Intervention): Those who received usual care

INTERVENTIONS:
Behavioral: Bone Mineral Density Result Letter and Bone Health Brochure — Letter mailed to patient to include - Date of DXA, T-score, impression, 10 year major fracture risk with visual depiction of risk, basic bone health guidelines, instructions to follow-up with their healthcare provider. The brochure will include information on osteoporosis, calcium, vitamin D, medicines, exercise, tobacco and alcohol cessation and where to find more information.
  Arms: BMD Result Letter and Brochure

SUMMARY:
There is growing evidence that patients undergoing bone mineral density testing (BMD) often do not take important steps to improve their bone health. The investigators will conduct a randomized-controlled trial to evaluate the impact of a novel and practical patient activation intervention (mailing patients their bone density test results) on the quality of bone-related healthcare and the cost-effectiveness of BMD testing. Equally important, the investigators intervention could easily be modified to include other patient populations and chronic diseases.

DETAILED DESCRIPTION:
Bone mineral density (BMD) peaks in early adulthood and declines progressively with aging. As BMD declines from normal, to low (formerly called osteopenia), to osteoporosis, risk of fractures progressively increases. In an effort to prevent bone loss and reduce fracture risk, most widely accepted guidelines including the U.S. Preventive Services Task Force and Surgeon General's Office now recommend BMD screening of older adults using dual energy x-ray absorptiometry (DXA). The rationale for screening is that patients and their providers will use DXA results as a "cue to action" and take necessary steps to enhance bone health through lifestyle modification (e.g., weight bearing exercise), Calcium/Vitamin D supplementation, and pharmacotherapy when indicated. However, multiple studies have demonstrated that patients and providers often fail take recommended actions following DXA testing, thus defeating much of the purpose of screening. Over the past five years we have systematically developed and pilot tested a low-cost and practical patient activation intervention based upon the Health Belief Model. The intervention consists of the DXA scanning center mailing each patient a customized letter containing the results of their DXA scan plus educational information about osteoporosis, supplemented by a follow-up phone call from a nurse educator. Preliminary studies have demonstrated that the intervention is well received by both patients and providers and enhances bone-related quality of care. The overarching objective of the current proposal is to rigorously examine the impact of our patient activation intervention on bone-related quality of care in adults undergoing screening DXA scans through a randomized-controlled trial conducted at three study sites. In addition, we will examine the real-world costs associated with our intervention and the impact of our intervention on the overall cost-effectiveness of BMD screening. We hypothesize that the activation intervention will increase optimization of Calcium/Vitamin D intake, enhance use of pharmacotherapy when indicated, will improve patient satisfaction with their bone-related healthcare, and improve patients' osteoporosis specific knowledge when compared with usual care

ELIGIBILITY:
Inclusion Criteria:

1. patients presenting for DXA
2. age 50 years of age or older

Exclusion Criteria:

1. non-English speakers
2. prisoners
3. people who have mental disabilities
4. individuals younger than age 50 years
5. individuals who do not have access to a telephone
6. deaf patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7749 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Wolinsky, PhD, Principal Investigator — University of Iowa
Locations (4):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente Georgia, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edmonds SW, Wolinsky FD, Christensen AJ, Lu X, Jones MP, Roblin DW, Saag KG, Cram P; PAADRN Investigators. The PAADRN study: a design for a randomized controlled practical clinical trial to improve bone health. Contemp Clin Trials. 2013 Jan;34(1):90-100. doi: 10.1016/j.cct.2012.10.002. Epub 2012 Oct 17. PMID 23085132
- [Background] Edmonds SW, Solimeo SL, Lu X, Roblin DW, Saag KG, Cram P. Developing a bone mineral density test result letter to send to patients: a mixed-methods study. Patient Prefer Adherence. 2014 Jun 5;8:827-41. doi: 10.2147/PPA.S60106. eCollection 2014. PMID 24940049
- [Background] Edmonds SW, Cram P, Lu X, Roblin DW, Wright NC, Saag KG, Solimeo SL; PAADRN Investigators. Improving bone mineral density reporting to patients with an illustration of personal fracture risk. BMC Med Inform Decis Mak. 2014 Nov 25;14:101. doi: 10.1186/s12911-014-0101-y. PMID 25743200
- [Background] Edmonds SW, Solimeo SL, Nguyen VT, Wright NC, Roblin DW, Saag KG, Cram P. Understanding Preferences for Osteoporosis Information to Develop an Osteoporosis Patient Education Brochure. Perm J. 2017;21:16-024. doi: 10.7812/TPP/16-024. Epub 2016 Nov 18. PMID 28080957
- [Result] Edmonds SW, Cram P, Lou Y, Jones MP, Roblin DW, Saag KG, Wright NC, Wolinsky FD; PAADRN Investigators. Effects of a DXA result letter on satisfaction, quality of life, and osteoporosis knowledge: a randomized controlled trial. BMC Musculoskelet Disord. 2016 Aug 26;17(1):369. doi: 10.1186/s12891-016-1227-0. PMID 27562713
- [Result] Wolinsky FD, Lou Y, Edmonds SW, Hall SF, Jones MP, Wright NC, Saag KG, Cram P, Roblin DW; PAADRN Investigators. Activating Patients With a Tailored Bone Density Test Results Letter and Educational Brochure: the PAADRN Randomized Controlled Trial. J Clin Densitom. 2017 Oct-Dec;20(4):464-471. doi: 10.1016/j.jocd.2016.08.012. Epub 2016 Sep 16. PMID 27647261
- [Result] Cram P, Wolinsky FD, Lou Y, Edmonds SW, Hall SF, Roblin DW, Wright NC, Jones MP, Saag KG; PAADRN Investigators. Patient-activation and guideline-concordant pharmacological treatment after bone density testing: the PAADRN randomized controlled trial. Osteoporos Int. 2016 Dec;27(12):3513-3524. doi: 10.1007/s00198-016-3681-9. Epub 2016 Jun 30. PMID 27363400
- [Derived] Roblin DW, Cram P, Lou Y, Edmonds SW, Hall SF, Jones MP, Saag KG, Wright NC, Cromwell LF, Robinson BE, Wolinsky FD; PAADRN Investigators. The Contribution of Patient, Primary Care Physician, and Primary Care Clinic Factors to Good Bone Health Care. Perm J. 2021 Jan;25:1-3. doi: 10.7812/TPP/20.095. PMID 33635767
- [Derived] Solimeo SL, Nguyen VT, Edmonds SW, Lou Y, Roblin DW, Saag KG, Cram P, Wolinsky FD. Sex differences in osteoporosis self-efficacy among community-residing older adults presenting for DXA. Osteoporos Int. 2019 May;30(5):1033-1041. doi: 10.1007/s00198-019-04854-6. Epub 2019 Jan 30. PMID 30701343
- [Derived] Hall SF, Wright NC, Wolinsky FD, Lou Y, Edmonds S, Roblin D, Jones M, Saag K, Cram P. The prevalence of overtreatment of osteoporosis: results from the PAADRN trial. Arch Osteoporos. 2018 Sep 28;13(1):103. doi: 10.1007/s11657-018-0517-6. PMID 30267162
- [Derived] Roblin DW, Cram P, Lou Y, Edmonds SW, Hall SF, Jones MP, Saag KG, Wright NC, Wolinsky FD; PAADRN Investigators. Diet and exercise changes following bone densitometry in the Patient Activation After DXA Result Notification (PAADRN) study. Arch Osteoporos. 2018 Jan 6;13(1):4. doi: 10.1007/s11657-017-0402-8. PMID 29307094
- [Derived] Wolinsky FD, Hall SF, Lou Y, Edmonds SW, Saag KG, Roblin DW, Wright NC, Jones MP, Cram P; PAADRN Investigators; Curtis JR, Morgan SL, Schlechte JA, Williams JH, Zelman DJ. The cost of a patient activation intervention for achieving successful outcomes: results from the PAADRN randomized controlled trial. Osteoporos Int. 2017 Oct;28(10):3061-3066. doi: 10.1007/s00198-017-4113-1. Epub 2017 Jun 15. PMID 28620779
- [Derived] Wolinsky FD, Lou Y, Edmonds SW, Saag KG, Roblin DW, Wright NC, Jones MP, Cram P; PAADRN Investigators. The effects of a patient activation intervention on smoking and excessive drinking cessations: results from the PAADRN randomized controlled trial. Osteoporos Int. 2017 Oct;28(10):3055-3060. doi: 10.1007/s00198-017-4101-5. Epub 2017 Jun 1. PMID 28573377
- [Derived] Cram P, Saag KG, Lou Y, Edmonds SW, Hall SF, Roblin DW, Wright NC, Jones MP, Wolinsky FD; PAADRN Investigators*. Racial Differences and Disparities in Osteoporosis-related Bone Health: Results From the PAADRN Randomized Controlled Trial. Med Care. 2017 Jun;55(6):561-568. doi: 10.1097/MLR.0000000000000718. PMID 28288074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting for DXA centers were recruited through February 2012 to August 2014 at three health centers-the University of Iowa (UI), the University of Alabama at Birmingham (UAB), and Kaiser Permanente of Georgia (KPGA).
Groups:
- Control: Usual care
Period: Overall Study
Arm/Group | BMD Result Letter and Brochure | Control
Started | 3898 | 3851
Completed | 3082 | 3020
Not Completed | 816 | 831
Not completed — Death | 26 | 18
Not completed — Withdrawal by Subject | 290 | 287
Not completed — Lost to Follow-up | 498 | 523
Not completed — Proxy interview done | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMD Result Letter and Brochure | Control | Total
Number analyzed (Participants) | 3898 | 3851 | 7749
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.4) | 66.7 (8.2) | 66.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3259 | 3230 | 6489
  Male | 639 | 621 | 1260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 77 | 151
  Not Hispanic or Latino | 3824 | 3774 | 7598
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 37 | 43 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 842 | 814 | 1656
  White | 2981 | 2954 | 5935
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 34 | 36 | 70
Region of Enrollment [Number; unit: participants]
  United States | 3898 | 3851 | 7749

OUTCOME MEASURES:

1. Primary Outcome: Guideline Concordant Osteoporosis Therapy
Description: Guideline concordant was defined as those who prescribed a National Osteoporosis Foundation approved osteoporosis therapy for patients with osteoporosis (T-score of femoral neck, hip, or spine ≤-2.5 or FRAX ≥20 %), or patients with a self-reported history of low impact fracture, or patients with osteopenia (T-score between -1.0 and -2.5 at the femoral neck, hips, or lumbar spine) and a 10-year probability of a major osteoporosis-related fracture ≥20 % OR those who were not prescribed a therapy for patients with no self-reported history of prior DXA and study DXA shows normal BMD and no self-reported history of low impact fracture, or study DXA shows osteopenia (T-score of femoral neck, hip, or spine between -1 and -2.5) and FRAX <20 %) and no self-reported history of low impact fracture, or self-reported prior DXA but no self-reported history of low impact fracture and no self-reported history of osteoporosis.
Time Frame: 12 weeks after DXA
Measure: Count of Participants; unit: Participants
Arm/Group | BMD Result Letter and Brochure | Control
Number analyzed (Participants) | 3898 | 3851
Participants | 2537 | 2477

ADVERSE EVENTS:
Time Frame: Due to the minimal risk nature of our study we did not collect adverse event data. We did track people for one year after enrollment.
Description: Due to the minimal risk nature of our study we did not collect adverse event data.
Arm/Group | BMD Result Letter and Brochure | Control
All-Cause Mortality (participants affected / at risk) | 26/3898 | 18/3851
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No